CLINICAL TRIAL: NCT03894592
Title: Utilizing Virtual Reality Analgesia (VRA) as a First Line Nonpharmacologic Analgesic Intervention on the Acute Rehabilitation Unit: A Pilot Study
Brief Title: Virtual Reality Analgesia In Trauma Rehab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-9196
Record Dates: First submitted 2018-10-29; First posted 2019-03-28 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Virtual Reality; Musculoskeletal Pain; Opioid Use; Anxiety; Virtual Reality Analgesia; Trauma Injury
MeSH Terms: conditions — Musculoskeletal Pain; Anxiety Disorders; Accidental Injuries

STUDY DESIGN:
Intervention Model Description: This is a Randomized control study. The pre and post VAS scores will be rated by the patient. Randomization will be achieved using Sequentially Numbered opaque sealed envelopes ( SNOSE) and an online randomization tool. All the patients will choose one of three virtual reality experiences.
  1. Passive VR Movie
  2. Interactive relaxation/exploration
  3. Active/Adventure experience
Who Masked: Investigator, Outcomes Assessor
Masking Description: Sequentially Numbered opaque sealed envelopes ( SNOSE) and an online randomization tool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality analgesia (Active Comparator): Trauma patients in rehab unit in the participating hospital will be included in this arm if they are randomized to receive the intervention which is a virtual reality headset providing immersive interactive content in the video format
  Interventions: Other: Virtual reality
- Control (No Intervention): Trauma patients in rehab unit in the participating hospital will be included in this arm if they are randomized to receive no intervention

INTERVENTIONS:
Other: Virtual reality — Trauma patients enrolled in the study will be offered Virtual Reality experieince per the protocol
  Arms: Virtual Reality analgesia

SUMMARY:
This will be a pilot study utilizing Virtual Reality Analgesia (VRA) as a first line nonpharmacologic analgesic intervention on the Acute Rehabilitation Unit. In order to assess the efficacy of the intervention with a set of outcome measures will be defined:

* Pain will be measured using the VAS for all subjects pre-, during and post-intervention via self-report.
* Number of opioids/oral pain medication consumed will be analyzed
* Patient anxiety will be measured on the Short ( State-Trait Anxiety Index) STAI anxiety scale pre- and post-intervention.
* Heart rate and blood pressure will also be measured pre and post intervention.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate the efficacy of virtual reality analgesia (VRA) for Adult patients in acute pain in the Acute Rehabilitation unit. Given the severity of the opioid epidemic, physicians are looking for alternative non-opioid/non-pharmacologic interventions to decrease both pain, and the need for opioids.

The recognition of pain by an individual requires both a noxious stimulus as well as attention on the part of the subject. Studies have shown that pain sensation is less on the visual analogue scale (VAS) when subjects are distracted, and that distraction can assist in pain control, since humans have limited attention capacity. When treating Adult patients with acute pain, it could thus be useful to have an effective method of pain distraction to improve tolerance and comfort, and to decrease the amount of narcotic medications prescribed.

Virtual reality (VR) is a digital simulation of a three-dimensional environment in which the user is capable of interacting with the generated world via computerized equipment such as gloves or a virtual reality head-mounted display (VRHMD). 360-degree VR video is a subset of virtual reality which creates an immersive experience of real world environments, allowing the user to have a sense of presence and exploration while wearing a (VRHMD). VR exposure is shown to be a potent distractor and has been repeatedly shown to provide analgesia during painful procedures. Since adults are often very attracted to technology, computer games, and virtual reality, we propose a study to allow adults to interact with a custom virtual reality environment in order to consume a substantial proportion of their attentional resources during acute pain episodes. We hypothesize that immersing the patients in VR will allow these patients to spend less attention on pain and allow for less need for other analgesia i.e. opioids.

VR has been demonstrated as a valid method of analgesia for both adults and pediatrics during painful procedures. To the investigator's knowledge, no one has evaluated the use of VRA to reduce opioid consumption in the Acute Rehab unit. In addition to relieving pain, anxiety, stress, and possibly decreasing general sedation, VRA may also decrease medical costs by decreasing length of stay.

Virtual Reality Analgesia (VRA) has been shown by research to be more effective when more immersive. To accomplish this, various head-sets and technologies have been developed to provide a more enveloping experience. Until recently, virtual reality head-mounted displays (VRHMD) had not been widely accepted due to their poor performance and high cost. But recent developments with the Oculus Rift DK1(DK 1 is a model number) in 2012 changed this paradigm. The now commercially available Oculus Rift is an inexpensive state of the art VRHMD. Using the Oculus Rift can create a high definition and smooth environment that will allow for maximal distraction at a modest price point. Therefore, equipment like the Oculus Rift could be an ideal VRA tool in the clinical setting.

Many corporations such as Samsung, Google, and others have invested both capital and development resources that have advanced virtual reality technologies and made them very inexpensive. With these changes, the investigators are finally at a point where both the hardware and the software needed to produce high quality VRHMD is now available at very low and moderate price points. An example of the lowest cost VRHMD is the Google Cardboard, a simple device that allows anyone with a cellphone to experience VR, for as little as $15.

The investigators propose a study utilizing the highest quality VRHMD to provide VRA during acute pain related to trauma. It is the investigators' hypothesis that by using VRA, significant decrease in the overall pain and discomfort can be observed resulting in a decrease in consumption of oral opioids.

ELIGIBILITY:
Inclusion Criteria:

* Adult with Traumatic injury on the Acute Rehab Unit
* Adult ages 18-100
* Adult with intact vision who can attend VR intervention
* Adult receiving PO Medications
* Adult with motor control of at least one arm

Exclusion Criteria:

* Adult who has uncontrolled seizures more than 4 times per year
* Adult who is not attentive to VR secondary to poor concentration/poor cognition to external stimuli.
* Adult with no volitional control of the neck and or upper extremities.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-07-02 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change in pain perception | 1 year
  will be measured using the Visual Analogue Scale (VAS) for all subjects pre-, during and post-intervention via self-report. The scale values range from 0 to 10. ) being no pain and 10 being the worst pain

SECONDARY OUTCOMES:
Increase or decrease in opioid/oral pain medication use | 1 year
  Number of opioids/oral pain medication consumed will be analyzed from the patients electronic medical record
Heart Rate | 1 year
  Pre and post intervention heart rate will be monitored using regular hospital equipment to note any changes pre and post intervention.
Patient reported anxiety | 1 year
  Anxiety will be measured on the Short STAI (State-Trait Anxiety Index) anxiety scale pre- and post-intervention.
  The scale has 2 parts with 20 questions in each part. Each question is rated on a 4 point scale,1 to 4.
  Total scores range from 20 to 80 for each part, with higher score indicating higher anxiety
Blood Pressure | 1 year
  Pre and post intervention blood pressure will be monitored using regular hospital equipment to note any changes pre and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Stern, MD, Principal Investigator — New York City Health and Hospitals Corporation
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No